CLINICAL TRIAL: NCT03914144
Title: Postnatal Prevalence of Bacteriuria in Women With Catheter Versus no Catheter in Labour: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/105/GHT
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Urinary Tract Infection in Pregnancy; Urinary Tract Infection Following Delivery; Catheter Infection
Keywords: catether; pregnancy; postnatal infection
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients are asked to provide 3 samples of urine which are to be processed in the laboratory with routine testing for microscopy, culture and sensitivity and disposed of in the standard way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Vaginal Delivery: The group of patients who achieved a normal delivery will be retrospectively assessed as to whether they had any episode of catheter insertion during their delivery.
  Interventions: Other: Catheter insertion
- Insturmental Vaginal Delivery: The group of patients who underwent instrumental delivery (ventouse or forceps) will be retrospectively assessed as to whether they had any episode of catheter insertion during their delivery.
  Interventions: Other: Catheter insertion
- Emergency Caesarean Section: Each patient will be recorded how many catheter episodes occurred during their labour and delivery.
  Interventions: Other: Catheter insertion
- Elective Caesarean Section: We expect all patients in this group to have an indwelling catheter sited before their elective caesarean sections, however we will assess each patient individually to confirm whether they had a catheter for their delivery.
  Interventions: Other: Catheter insertion

INTERVENTIONS:
Other: Catheter insertion — A data collection sheet will be assigned for every patient who is recruited for the study. The clinician caring for the patient will be asked to fill in this form after the delivery has occurred. The form essentially will describe if the patient received any catheter during the delivery and if so, an indwelling catheter or an intermittent (in/out) catheter and how many episodes this occurred.

SUMMARY:
Catheterisation is an accepted tool in intrapartum bladder care and indwelling catheters are used routinely before elective caesarean sections. However, urinary catheters are associated with an increased rate of urinary tract infections which can lead to complications including increased maternal morbidity and prolonged hospital stay. A Cochrane Review (2014) concluded that there is insufficient evidence to assess the routine use of indwelling bladder catheters in women undergoing caesarean section. The incidence and causation of catheter-associated infection in this population is unknown. We propose to provide this data, by comparing urine samples from pregnant women before and after their delivery and analysing this against observational catheter use during the delivery. This will be vital in conducting future research into potential change in policy on routine catheterisation. It will also be beneficial to patients as it could reduce the burden of catheterisation by reducing their chance of developing a UTI and by reducing the associated morbidity.

DETAILED DESCRIPTION:
Research Question

Is the intrapartum use of a catheter - either intermittent or indwelling - associated with an increased incidence of postnatal bacteriuria when compared with women who are not catheterised?

Method

Pregnant women will be recruited at Gloucestershire Royal Hospital Maternity Department from 37 weeks gestation. Once eligibility is met, they will be asked to provide a mid-stream urine sample which will be tested for microscopy, culture and sensitivity (MC&S). They will be analysed according to their mode of delivery. Their notes will be scrutinised to assess whether or not a catheter was sited during their labour. Postnatally, they will be asked to provide an MSU on day 3 and day 28, which will both be sent for MC&S. A comparative analysis between each MSU will be performed and correlated to whether intrapartum catheterisation was undertaken.

Data Collection & Analysis

The data collection phase will take approximately three months, with data analysis and write-up estimated to take a further one-two months.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study

  * Intact membranes
  * At least 37 weeks pregnant

Exclusion Criteria:

* • History of microbiologically-confirmed bacteriuria in preceding 28 days

  * Patients who are in active labour
  * Women who have had either urine-specific or broad-spectrum antibiotics within the last 28 days

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The target of recruitment is pregnant women from 37 weeks gestation. They will be recruited from the Maternity Triage Department, Antenatal Clinic, Central Delivery Suite, Birth Unit or the Maternity Ward.
Sampling Method: Probability Sample
Enrollment: 638 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Urinary Tract Infection | 30 days post delivery
  Postpartum urinary tract infection within 30 days of delivery, defined as positive MSU (>107 cfu/l) with associated symptoms.

SECONDARY OUTCOMES:
Postpartum asymptomatic bacteriuria | 30 days post delivery
  Postpartum asymptomatic bacteriuria detected within 30 days of delivery, defined as positive MSU (>107 cfu/l) without associated symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark James, MbChb, Principal Investigator — Gloucestershire NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
Patient information will be kept confidentially and not shared as per the Data Protection Act 2018